CLINICAL TRIAL: NCT02770014
Title: Rapid Plasma Genotyping For Early Initiation Of Erlotinib In EGFR Mutant Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to Osimertinib approval
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Principal Investigator, Geoffrey Oxnard, MD, Geoffrey Oxnard, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-093
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Epidermal Growth Factor Receptor; Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Epidermal Growth Factor Receptor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGFR mutation Positive, Treatment With Erlotinib (Experimental): Eligible EGFR mutations include exon 19 deletion or exon 21 L858R mutation. Erlotinib will be initially dosed at a pre-determine dosage daily, and it will be given on a 6-week cycle with treatment administered on an outpatient basis
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib
  Other Names: Tarceva

SUMMARY:
Patient with Non-Small Cell Lung Cancer (NSCLC) that might have a genetic change (mutation) in the Epidermal Growth Factor Receptor (EGFR) are invited to take part in this study.

This research study is evaluating a new blood test that is capable of detecting an EGFR mutation in cancer without a biopsy.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. This research study will determine if a rapid blood test can be used to detect EGFR mutations in patients with newly diagnosed lung cancer and use that information to rapidly start patients on a pill-based therapy.

This blood test has not previously been used to select patients for treatment with Erlotinib without confirming this finding on a biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic NSCLC including recurrent disease
* EGFR genotype must not be known. However, pending EGFR tumor genotyping is allowed.

  --Participants with positive or pending EGFR mutation on plasma genotyping performed at the central lab are eligible for enrollment, and will not need to repeat initial plasma genotyping on study.
* Tissue must be available for genotyping or biopsy planned to obtain tissue for genotyping. Biopsy requirement may be waived if not technically feasible and plasma genotyping reveals an eligible EGFR mutation (exon 19 del/L858R). Determination of technical feasibility must be made independently of plasma genotyping results.
* Participants must possess at least two of the following clinical characteristics which enrich for EGFR mutations:

  * smoked less than 10 pack years
  * Asian race.
  * Adenocarcinoma (including adenosquamous carcinoma) on histology or cytology.
* Participants must have measurable disease with at least one lesion that can be accurately measured in longest dimension as >2 cm with conventional imaging techniques or >1 cm with a spiral CT scan per RECIST v1.1.
* Participants must have progressive, advanced cancer as defined by one of the following:

  * Newly diagnosed, untreated advanced disease
  * Newly diagnosed, untreated metastatic recurrence of earlier stage disease (previous treatment of early stage disease allowed).
  * Clinical determination of progressive disease on previous systemic therapy as evidenced by plan to change treatment. Any number of prior therapies are acceptable excluding previous EGFR kinase inhibitors.
* Age 18 years or older.
* ECOG performance status 0-2.
* Participant must be able to understand and give consent to participate in the study.
* Patient must be a candidate for systemic therapy with erlotinib based on clinical assessment. Patients must meet the following criteria before beginning therapy (Note: these are not required for initial study enrollment and plasma genotyping):

  * ECOG performance status of 0-2
  * Platelets >75
  * AST & ALT < 3x the upper limit of normal
  * Creatinine clearance > 30 mL/min by Cockroft-Gault
  * No other contraindication to erlotinib
  * Female participants of child-bearing age must agree to use adequate contraception (hormonal, barrier or abstinence) for the duration of the study while receiving erlotinib and undergo a pregnancy test. Any evidence or suspicion of pregnancy should be reported to the treating physician immediately.
  * Male participants must agree to use adequate contraception for the duration of the study while receiving erlotinib

Exclusion Criteria:

* Participants must not have had chemotherapy within the past 10 days.
* Participants must not have had prior treatment with an EGFR kinase inhibitor, EGFR directed therapy or investigational agent.
* Participants must not have residual adverse events from previous therapy greater than CTCAE v4.0 grade 2 at the time of registration.
* Participants must not have symptomatic brain metastases or brain metastases requiring steroids. Asymptomatic brain metastases not requiring steroids are acceptable.
* Participant must not have a history of allergy to erlotinib.
* Second primary cancer which is active and requiring treatment.
* Participants must not be pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06; Primary Completion 2019-04-16 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey R Oxnard, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Plasma Genotyping: Participants who enrolled to the study and had plasma genotyping
Period: Plasma Genotyping
Arm/Group | Participants With Plasma Genotyping
Started | 43
Completed | 43
Not Completed | 0
Period: EGFR Exon 19 Pos, Treated With Erlotinib
Arm/Group | Participants With Plasma Genotyping
Started | 11 (A total of 11 participants were found to have an activating EGFR mutation (exon 19 del or L858R).)
Completed | 6 (Of the 11 participants that had an activating EGFR mutation, 6 started erlotinib treatment.)
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: All participants who enrolled to the study and had plasma genotyping performed
Arm/Group | Participants With Plasma Genotyping
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: years] | 63 [32 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 43
Smoking Status [Count of Participants; unit: Participants]
  Former Smoker | 14
  Never Smoker | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Number of participants who were alive with evidence of complete or partial response, evaluated using RECIST 1.1 criteria. Patients that underwent rapid plasma genotyping and had an EGFR mutation and who were treated with erlotinib were included in this calculation.
Time Frame: From date of erlotinib initiation until the date of first documented disease progression or date of death from any cause, whichever came first. ORR was assessed up to 21 months after erlotinib initiation.
Population: A total of 6 participants were treated with erlotinib on study.
Measure: Count of Participants; unit: Participants
Groups:
- EGFR Exon 19 Positive Treatment With Erlotinib: Erlotinib will be initially dosed at a pre-determine dosage daily, and it will be given on a 6-week cycle with treatment administered on an outpatient basis
Arm/Group | EGFR Exon 19 Positive Treatment With Erlotinib
Number analyzed (Participants) | 6
Participants | 4

2. Secondary Outcome: Turnaround Time
Description: The turnaround time from study registration to treatment initiation was recorded for the plasma genotyping strategy versus standard tumor genotyping. For rapid plasma genotyping, turnaround time is the time between ordering plasma genotyping and obtaining results; this time period was compared to the turnaround time of obtaining the tumor genotyping results.
Time Frame: Maximum 38 days
Population: A total of 42 participants had plasma genotyping results available (1 of the 43 enrolled participants did not have plasma genotyping).
Measure: Median (Full Range); unit: days
Arm/Group | Participants With Plasma Genotyping
Number analyzed (Participants) | 42
days
  Turnaround Time: Plasma Genotyping | 4 [1 to 11]
  Turnaround Time: Tumor Genotyping: number analyzed (Participants) | 35
  Turnaround Time: Tumor Genotyping | 20 [8 to 38]

3. Secondary Outcome: Positive Predictive Value (PPV) And False Negative Rate Of Plasma Genotyping
Description: Concordance between results of plasma genotyping and tumor genotyping, among patients with tissue available for standard genotyping
Time Frame: PPV and False Negative Rate can be assessed when plasma and tissue results are available for each patient; average plasma result turnaround time was 4 days, versus average of 20 days for tissue result turnaround time.
Population: 35 of the 42 participants with plasma genotyping results also had tumor genotyping results available, so PPV and false negative rate could be assessed in these 35 participants.
Measure: Number; unit: percentage
Arm/Group | Participants With Plasma Genotyping
Number analyzed (Participants) | 35
percentage
  Positive Predictive Value | 100
  False Negative Rate | 30

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the 6 participants who received erlotinib treatment from time of initiation of erlotinib through end of study. This time frame was a maximum of 21 months from initiation of erlotinib treatment to study completion.
Description: CTCAE version 4.03 was used for reporting adverse events. Serious Adverse Events were not collected/assessed for the Plasma Genotyping Participants, unless felt to be related to the study procedures. No such SAEs occurred on this study.
Arm/Group | EGFR Exon 19 Positive Treatment With Erlotinib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGFR Exon 19 Positive Treatment With Erlotinib (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (5)
Pain (General disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Paronychia (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (4)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin/subcutaneous tissue disorders; Other, specify (Skin and subcutaneous tissue disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/14/NCT02770014/Prot_SAP_000.pdf